CLINICAL TRIAL: NCT06424652
Title: Effect of Physiologic Insulin Administration on Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Frank Greenway, Professor-Chief Medical Officer, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBRC 2024-014
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Blood Specimen Collection; Basal Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Participant with Evidence of cognitive impairment. (Other)
  Interventions: Other: Blood draws; Other: Hyperinsulinemic Euglycemic Clamp Technique Insulin Sensitivity test; Other: Resting Metabolic Rate (RMR)

INTERVENTIONS:
Other: Blood draws — After passing the screening, participation in the research study will be approximately three weeks. The participant will have seven study visits all at the Pennington Center. On five occasions, the participant will have a five-hour visit in the inpatient unit. At the study visit blood will be drawn. The total amount of blood drawn during the study is approximately 12 fluid ounces.
Other: Hyperinsulinemic Euglycemic Clamp Technique Insulin Sensitivity test — This procedure measures how the body responds to insulin. Insulin is normally produced by the body during meals and helps the body use sugar. There will be two IV lines, one in the participant's arm and one in the participant's hand on the opposite side. Small amounts of glucose and insulin will be infused into the participant's arm. The participant's blood sugar level will be checked every 5-10 minutes from the IV in the hand to determine how much glucose the participant should have to keep blood sugar at a normal level. The participant's hand will be placed inside a warming box to increase skin temperature to about 105 degrees Fahrenheit. The temperature will be warm, but not uncomfortable. During the IV procedure, a small amount of the participant's own blood (less than 1 teaspoon) will immediately be returned into the vein through the IV after each specimen is collected.
Other: Resting Metabolic Rate (RMR) — After the participant rests for 30 minutes, a clear plastic hood will be placed over the participant's head and chest area. The hood is ventilated with fresh air. The participant's oxygen intake and carbon dioxide output will be measured for 30 minutes to determine how many calories the participant burns during the time they are being tested.

SUMMARY:
In humans, insulin is secreted in pulses from the pancreatic beta-cells, and these oscillations help to maintain fasting plasma glucose levels within a narrow normal range. These pulses become disrupted in the presence of insulin resistance. Some people have referred to Alzheimer's Disease as type 3 diabetes because the glucose uptake in the brain is reduced by 30%. Clinical observations in clinics that treat patients with insulin pulses every 5 minutes for 3 hours twice a week for 2 weeks followed by once a week for 6 weeks and followed by less frequency treatments suggest an improvement in type 2 diabetes control, reduction in insulin resistance and an improvement in diabetes complications. A patient with Parkinson's Disease was treated with this pulsed insulin paradigm and experienced dramatic improvement that has now been maintained over years. Parkinson's Disease has been reported to have a decreased glucose uptake in the brain, so pulsed insulin treatment was tried in a small number of patients with Alzheimer's Disease and there was an impression that they showed improvement. Clinics that use pulsed insulin treatment change more than one parameter of the insulin pulses which makes it difficult to determine what is giving the improvement. The euglycemic hyper-insulinemic clamp, also called a clamp, is a well-standardized test that measures insulin resistance and involves intravenous insulin infusion. This single patient study will enroll one patient with early Alzheimer's disease and insulin resistance. The subject will have one standard clamp test with continuous insulin followed by 4 clamps over a 2-week period using the same amount of insulin over the same period of time but administered in pulses every 5 minutes. This was the number of pulsed insulin treatments needed to see a dramatic improvement in Parkinson's disease. The cognition in the Alzheimer's disease patient will be thoroughly evaluated with questionnaires and walking on a special mat while doing arithmetic tasks before and after the 4 pulsed insulin clamps. If this study demonstrates an improvement in cognition, one will know that the only thing that changed from the standard clamp was the pulse nature of the insulin delivery.

DETAILED DESCRIPTION:
The purpose of this research study is to test the effect of an insulin treatment on Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Early Alzheimer's Disease
* Insulin Resistance

Exclusion Criteria:

* Inability to walk
* Unable to read, understand or inability to complete questionnaire
* Belong to a vulnerable group like prisoners

Ages: 65 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Effect of tissue sensitivity to insulin | Two weeks
  To determine the effect of tissue sensitivity to insulin delivered in pulses compared to insulin delivered continuously during the hyperinsulinemic euglycemic clamp test (clamp). The hypothesis is that delivery of insulin in pulses during the clamp (pulsatile clamp) will increase glucose disposal rate (GDR) compared to continuous delivery during the clamp (continuous clamp). To test the hypothesis, we will measure GDR during one pulsatile clamp and one continuous clamp at 40mU/m2/min insulin infusion.

SECONDARY OUTCOMES:
Effect of the pulsatile clamp at 40mU/m2/min insulin infusion on signs and symptoms of Alzheimer's disease | Two weeks
  To determine the effect of the pulsatile clamp at 40mU/m2/min insulin infusion on signs and symptoms of Alzheimer's disease. The hypothesis is that the signs and symptoms of Alzheimer's disease will improve following four pulsatile clamp treatments. To test the hypothesis, we will conduct assessments of cognition, homeostatic model assessment of insulin resistance, and brain insulin resistance prior to and following four pulsatile insulin clamps conducted twice weekly for two weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Penningto Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Protocol of the Nutrition Obesity Reseach Center - An NIH Center grant to Pennington and other National sites.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: July 1, 2025
Access Criteria: According to the Nutrition Obesity Research Center Protocol for sharing
URL: https://www.norc.org/

REFERENCES:
- [Result] Mergenthaler P, Lindauer U, Dienel GA, Meisel A. Sugar for the brain: the role of glucose in physiological and pathological brain function. Trends Neurosci. 2013 Oct;36(10):587-97. doi: 10.1016/j.tins.2013.07.001. Epub 2013 Aug 20. PMID 23968694
- [Result] Leclerc M, Bourassa P, Tremblay C, Caron V, Sugere C, Emond V, Bennett DA, Calon F. Cerebrovascular insulin receptors are defective in Alzheimer's disease. Brain. 2023 Jan 5;146(1):75-90. doi: 10.1093/brain/awac309. PMID 36280236
- [Result] Cull O, Al Qadi L, Stadler J, Martin M, El Helou A, Wagner J, Maillet D, Chamard-Witkowski L. Radiological markers of neurological manifestations of post-acute sequelae of SARS-CoV-2 infection: a mini-review. Front Neurol. 2023 Nov 24;14:1233079. doi: 10.3389/fneur.2023.1233079. eCollection 2023. PMID 38073629
- [Result] Chun MY, Chung SJ, Kim SH, Park CW, Jeong SH, Lee HS, Lee PH, Sohn YH, Jeong Y, Kim YJ. Hippocampal Perfusion Affects Motor and Cognitive Functions in Parkinson Disease: An Early Phase 18 F-FP-CIT Positron Emission Tomography Study. Ann Neurol. 2024 Feb;95(2):388-399. doi: 10.1002/ana.26827. Epub 2023 Nov 28. PMID 37962393
- [Result] Zhang Q, Fan C, Wang L, Li T, Wang M, Han Y, Jiang J; Alzheimer's Disease Neuroimaging Initiative. Glucose metabolism in posterior cingulate cortex has supplementary value to predict the progression of cognitively unimpaired to dementia due to Alzheimer's disease: an exploratory study of 18F-FDG-PET. Geroscience. 2024 Feb;46(1):1407-1420. doi: 10.1007/s11357-023-00897-0. Epub 2023 Aug 23. PMID 37610594
- [Result] Kapogiannis D, Boxer A, Schwartz JB, Abner EL, Biragyn A, Masharani U, Frassetto L, Petersen RC, Miller BL, Goetzl EJ. Dysfunctionally phosphorylated type 1 insulin receptor substrate in neural-derived blood exosomes of preclinical Alzheimer's disease. FASEB J. 2015 Feb;29(2):589-96. doi: 10.1096/fj.14-262048. Epub 2014 Oct 23. PMID 25342129
- [Result] Tam CS, Xie W, Johnson WD, Cefalu WT, Redman LM, Ravussin E. Defining insulin resistance from hyperinsulinemic-euglycemic clamps. Diabetes Care. 2012 Jul;35(7):1605-10. doi: 10.2337/dc11-2339. Epub 2012 Apr 17. PMID 22511259
- [Result] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Result] Lin JS, O'Connor E, Rossom RC, Perdue LA, Burda BU, Thompson M, Eckstrom E. Screening for Cognitive Impairment in Older Adults: An Evidence Update for the U.S. Preventive Services Task Force [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2013 Nov. Report No.: 14-05198-EF-1. Available from http://www.ncbi.nlm.nih.gov/books/NBK174643/ PMID 24354019
- [Result] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Result] Feng YS, Kohlmann T, Janssen MF, Buchholz I. Psychometric properties of the EQ-5D-5L: a systematic review of the literature. Qual Life Res. 2021 Mar;30(3):647-673. doi: 10.1007/s11136-020-02688-y. Epub 2020 Dec 7. PMID 33284428